CLINICAL TRIAL: NCT05124977
Title: Antimicrobial Stewardship For Ventilator Associated Pneumonia in Intensive Care
Acronym: ASPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: APHP200011
Record Dates: First submitted 2021-11-15; First posted 2021-11-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Antimicrobial Stewardship

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Antimicrobial stewardship based on daily clinical assessment of clinical cure (experimental group). Discontinuation of antibiotic therapy antibiotics if criterions of clinical cure (regression of tracheal secretions, regression of temperature, improvement of PaO2/FiO2 ratio, absence of hemodynamic failure) of confirmed VAP are met. In the intervention group, intensivists will perform clinical assessment daily in order to decide on the pursuit or discontinuation of antibiotic therapy.
  Interventions: Drug: Antimicrobial Stewardship
- Control group (Other): Standard management: duration of appropriate antibiotic therapy for confirmed VAP according to guidelines. In the control group, intensivists will perform clinical assessment daily, but a minimum duration of 7 days, as highly recommended of antibiotic therapy will be mandatory whatever the clinical cure.
  Interventions: Drug: Standard management

INTERVENTIONS:
Drug: Antimicrobial Stewardship — Antimicrobial stewardship based on daily clinical assessment of clinical cure. Discontinuation of appropriate antibiotic therapy antibiotics if criteria of clinical cure of confirmed pneumonia are met. Intensivists will perform clinical assessment daily in order to decide on the pursuit or discontinuation of antibiotic therapy.
  Arms: Experimental group
Drug: Standard management — Standard management: duration of appropriate antibiotic for confirmed pneumonia fixed for 7 days according to guidelines. In the control group, intensivists will perform clinical assessment daily, but the antibiotic will not be discontinued until 7 days whatever the clinical cure.
  Arms: Control group

SUMMARY:
Increasing emergence of multidrug resistant (MDR) bacteria worldwide is now considered one of the most urgent threats to global health. The association between increase of antibiotics consumption and resistance emergence has been well documented for all patients admitted to the Intensive care unit (ICU) who received antibiotic treatment and for patients treated for ventilator associated pneumonia (VAP).

Reduction of use of antibiotics is a major point in the war against antimicrobial resistance. VAP is the first cause of healthcare-associated infections in ICU and more than half of antibiotics prescriptions in ICU are due to VAP.

Once the diagnosis of pneumonia under MV has been made, initiation of antibiotic treatment must be prompt but there is no clear consensus on its duration. In the case of a good clinical response to treatment, it has been shown in some situations that short course antibiotics can be effective without side effects and antimicrobial stewardship initiatives can be applied successfully and effectively to the management of Community Acquired Pneumonia (CAP).

The hypothesis is that an antimicrobial stewardship is possible in the treatment of VAP with no increase in the rate of all-cause mortality, treatment failure or occurrence of new episode of pneumonia.

The objective is to investigate whether an antimicrobial stewardship for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in terms of all-cause mortality, treatment failure or occurrence of new episode of pneumonia.

This study will be a prospective, national multicenter (31 centers), phase III, comparative randomized (1:1), single-blinded clinical trial comparing two management strategies of treatment of pneumonia on the basis of two parallel arms:

Experimental group: Antimicrobial stewardship based on daily clinical assessment of clinical cure.

Control group: standard management: duration of appropriate antibiotic therapy for confirmed VAP according to guidelines.

DETAILED DESCRIPTION:
Increasing emergence of multidrug resistant (MDR) bacteria worldwide is now considered one of the most urgent threats to global health. The association between increase of antibiotics consumption and resistance emergence has been well documented for all patients admitted to the Intensive care unit (ICU) who received antibiotic treatment1 and for patients treated for ventilator associated pneumonia (VAP). Reduction of use of antibiotics is a major point in the war against antimicrobial resistance. VAP is the first cause of healthcare-associated infections in ICU and more than half of antibiotics prescriptions in ICU are due to VAP. Current international guidelines define VAP as a pneumonia occurring>48 hours after endotracheal intubation and distinguishes early onset VAP occurring in the first five days after admission and late VAP, occurring after.

Once the diagnosis of pneumonia under MV has been made, initiation of antibiotic treatment must be prompt but there is no clear consensus on its duration. In the case of a good clinical response to treatment, it has been shown in some situations that short course antibiotics can be effective without side effects and antimicrobial stewardship initiatives can be applied successfully and effectively to the management of Community Acquired Pneumonia (CAP).

American guidelines strongly recommend a 7-day course of antibiotic therapy rather than a longer duration but remark that "there exist situations in which a shorter or longer duration of antibiotics may be indicated, depending upon the rate of improvement of clinical, radiologic, and laboratory parameters".

The hypothesis is that an antimicrobial stewardship is possible in the treatment of VAP with no increase in the rate of all-cause mortality, treatment failure or occurrence of new episode of pneumonia.

The objective is to investigate whether an antimicrobial stewardship for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in terms of all-cause mortality, treatment failure or occurrence of new episode of pneumonia.

This study will be a prospective, national multicenter (31 centers), phase III, comparative randomized (1:1), single-blinded clinical trial comparing two management strategies of treatment of pneumonia on the basis of two parallel arms:

Experimental group: Antimicrobial stewardship based on daily clinical assessment of clinical cure.

Control group: standard management: duration of appropriate antibiotic therapy for confirmed VAP according to guidelines.

The primary endpoint is a hierarchical endpoint with a first non-inferiority criteria and a second efficacy criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of microbiologically confirmed of first episode of VAP
* Initial appropriate antibiotic therapy (whether empirical or not)
* Written informed consent from the patient or a legal representative if appropriate. If absence of a legal representative the patient may be included in emergency procedure

Definitive diagnosis of pneumonia (in agreement with international guidelines) is defined by association:

* Patient under MV>48 hours at the time of the microbiological sampling
* New pulmonary infiltrate of which an infectious origin is strongly suspected
* Worsening oxygenation
* Have the following clinical criteria within the 24 hours prior to the first dose of antibiotic therapy

  * Purulent tracheal secretions
  * And at least 1 of the following : documented fever (body temperature >38,3°C) or hypothermia (body temperature <35°C) or white blood cell (WBC) count >10,000 cells/mm3 or <4,000 cells/mm3
* Microbiological criteria (positive quantitative culture of a lower respiratory tract (LRT): bronchoalveolar lavage fluid (BAL) (significant threshold ≥10^4 colony-forming units/mL) or plugged telescopic catheter (PTC) (significant threshold ≥ 10^3 colony-forming units/mL) or quantitative endotracheal aspirate (ETA) distal pulmonary secretion samples (significant threshold ≥10^5 colony-forming units/mL)

Exclusion Criteria:

* Patient under selective decontamination of the digestive tract
* Duration of antibiotic therapy prior to inclusion > 72h (for any reason) appropriate to the germs found in the bacterial documentation of the first episode of VAP
* Inclusion in another interventional study concerning antimicrobial strategies
* Moribund (IGS II>80)
* Thoracic trauma with Abbreviated Injury Scale (AIS) thorax ≥ 3
* Severely immunocompromised patients (such as congenital immunodeficiency, neutropenia (<1leucocyte/ml or <0.5 neutrophil/ml) or acute hematologic malignancy or stem cell transplant, HIV infection with CD4 count below 200/mm3
* Patients undergoing immunosuppressive therapy and long term corticotherapy > 0.5 mg/kg
* VAP due to: Pseudomonas aeruginosa, Carbapenem-resistant Acinetobacter spp, Carbapenem-resistant Enterobacteriaceae
* VAP occurring in the context of co-infection of COVID-19 or other viral pneumonia (confirmed by RT-PCR)
* Patients with empyema, necrotizing and abscessed pneumonia
* Patients requiring extracorporeal oxygen therapy (ECMO), either veno-venous or veno-arterial
* Pregnant women
* No health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in terms of all-cause mortality, treatment failure or occurrence of new episode of pneumonia | 28 days
  The primary endpoint is a composite endpoint with non-inferiority criteria including:
  1. all-cause mortality (ACM) measured at day 28 after initiation of therapy
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in terms of all-cause mortality, treatment failure or occurrence of new episode of pneumonia | 28 days
  The primary endpoint is a composite endpoint with non-inferiority criteria including:
  2. Treatment failure defined by new signs of pneumonia within 72 hours after the end antibiotic treatment at the test of cure visit
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in terms of all-cause mortality, treatment failure or occurrence of new episode of pneumonia | 28 days
  The primary endpoint is a composite endpoint with non-inferiority criteria including:
  3. New episode of microbiologically confirmed VAP from 72H after the end of antibiotic treatment to day 28 after initiation of VAP antibiotic treatment

SECONDARY OUTCOMES:
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in term of all-cause mortality | 28 days after inclusion
  Rate of all-cause mortality
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in term of occurrence of treatment failure | 28 days after inclusion
  Rate of treatment failure
investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would be non-inferior in term of occurrence of new episode of pneumonia | 28 days after inclusion
  Rate of new episode of VAP
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would increase the number of antibiotic free-alive days, from initiation of VAP antibiotic therapy to day 28 | 28 days after inclusion
  Number of antibiotic free alive-days
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would reduce at day 28 after inclusion of VAP antibiotic therapy the global DOOR score | 28 days after inclusion
  Global score constructed with the DOOR and RADAR
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would reduce at day 28 after inclusion the duration of invasive mechanical ventilation | 28 days after inclusion
  Duration of invasive MV
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would reduce at day 28 after inclusion the length of stay in intensive care unit | 28 days after inclusion
  Length of ICU stay
To investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would reduce at day 28 after inclusion the rate of VAP recurrence | 28 days after inclusion
  Rate of VAP recurrence
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would reduce at day 28 after inclusion the rate of complications of antibiotic therapy | 28 days after inclusion
  Rate of antibiotic related side effects
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would reduce at day 28 after inclusion the rate of acquisition of carriage of MDR bacteria | 28 days after inclusion
  Rate of acquisition of MDR bacteria
Investigate whether an AMS for VAP based on daily assessment of clinical cure and antimicrobial discontinuation, if it is obtained, would reduce at day 28 after inclusion: The rate of subsequent infection due to : carbapenem-resistant Enterobacteriaceae | 28 days after inclusion
  Rate of subsequent infection of MDR bacteria
Study if an AMS based on daily clinical assessment of clinical cure of VAP versus standard management would improve survival at days 28 and 90 after inclusion | 28 and 90 days after inclusion
  Rate of death
Study the adherence to the AMS strategy (in order to identify factors associated to this adherence) in the intervention group only at day 28 after inclusion | 28 days after inclusion
  Adherence to AMS strategy
Assess the medico-economic impact of antimicrobial stewardship applied to VAP at day 28 after inclusion | 28 days after inclusion
  Total cumulative costs

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Foucrier, Principal Investigator — APHP
Locations (1):
- Foucrier, Clichy-sous-Bois, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Foucrier A, Roquilly A, Bachelet D, Martin-Loeches I, Bougle A, Timsit JF, Montravers P, Zahar JR, Eloy P, Weiss E; ASPIC study group. Antimicrobial Stewardship for Ventilator Associated Pneumonia in Intensive Care (the ASPIC trial): study protocol for a randomised controlled trial. BMJ Open. 2023 Feb 21;13(2):e065293. doi: 10.1136/bmjopen-2022-065293. PMID 36810173